## **ENGLISH CONSENT FORM**

The study you are about to participate is a randomized control trial survey titled as;

"Effects of Supervised Structured Aerobic Exercise training program on serum BDNF, androgens level, menstrual irregularity and quality of life in females with Insulin resistant polycystic ovarian syndrome."

The study has no potential harm to participants. All data collected from you will be coded in order to protect your identity, and should not be disclosed to anyone. Following the study there will be no way to connect your name with your data. Your answers to the questions will not affect the quality of education given to you. Any additional information about the study results will be provided to you at its conclusion, upon your request.

You are free to withdraw from the study at any time. You agree to participate, indicating that you have read and understood the nature of the study, and that all your inquiries concerning the activities have been answered to your satisfaction.

| NAME | SIGNATURE |
|------|-----------|
| DATE | |